CLINICAL TRIAL: NCT00661518
Title: Imaging of Aneurysm Wall Inflammation Using Positron Emission Tomography.
Brief Title: PET/CT Imaging of Aneurysm Wall Inflammation
Acronym: ASAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: M. Truijers, MD, Radboud University Nijmegen Medical Centre
Other Study IDs: ASAP
Record Dates: First submitted 2008-04-14; First posted 2008-04-18 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2008-04

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients scheduled for conventional aneurysm repair
- 2: Patients scheduled for endovascular aneurysm repair

SUMMARY:
Rationale: Aneurysm development, progression and rupture are characterised by extensive inflammation, dominated by the infiltration of T-cells, B-cells and macrophages. Recent studies into the pathophysiology of aneurysm wall degradation suggest a close relation between increased mechanical stress and the local activation of infiltrated lymphocytes and macrophages. The non-invasive detection of aneurysm wall inflammation, using 18-fluorodeoxyglucose positron emission tomography (FDG-PET) might therefore provide valuable information on the extend of the disease and could clarify the role of mechanical stress on the propagation of aneurysm wall inflammation.

Objective: Correlation of FDG uptake and in vitro aneurysm wall tensile strength. (primary objective). The effect of aneurysm sac depressurisation, after endovascular aneurysm repair, on aneurysm wall inflammation (secondary objective).

Study design: Observational case series (pilot). Study population: Patients scheduled for conventional (open) and endovascular aneurysm repair.

Main study parameters: Standard uptake value (SUV) measurements to asses FDG uptake in the aneurysm wall and in vitro aneurysm wall strength (N/mm).

Nature and extent of the burden and risks associated with participation,

benefit and group relatedness: Patients scheduled for conventional (open) or endovascular aneurysm repair are admitted to the hospital the day before surgery. At that point all patients will be evaluated using FDG-PET. Although intake of sugar-free liquids is permitted, glucose intake is restricted 6 hours prior to FDG-PET imaging. One hour after intravenous injection of 200-220 MBq FDG, whole body emission and transmission images will be acquired. To determine inflammation markers ( e.g. CRP), blood and urine samples will be collected prior to the operation and again 6 weeks after surgery. For in vitro aneurysm wall tensile strength testing wall specimens will be harvested during conventional aneurysm repair.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for conventional (10 patients) or endovascular (25 patients) aneurysm repair.
* Informed consent

Exclusion Criteria:

* Diabetes Mellitus type 1 en 2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population: At the Radboud University Nijmegen Medical Centre, approximately 80 patients undergo prophylactic aneurysm repair each year. 10-15 patients are scheduled for conventional ('open') repair the remaining 65-70 patients undergo endovascular aneurysm. We therefore expect to finish including patients for both studies by the end of august 2008. The study population will be comprised both male (± 80%) and female patients with an abdominal aortic aneurysm.
  Inclusion criteria
  Exclusion criteria
  -Diabetes Mellitus type 1 en 2
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-10 (Estimated); Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Truijers, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands